CLINICAL TRIAL: NCT04396379
Title: ENRAPTUS Epicardial Mitral Touch System for Mitral Insufficiency
Brief Title: Epicardial Mitral Touch System for Mitral Insufficiency
Acronym: ENRAPTUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mitre Medical Corp. (Industry)
Collaborators: BSWRI Cardiac Imaging Core Lab (CICL) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: TPL0002
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Ischemic Mitral Regurgitation; Functional Mitral Regurgitation

STUDY DESIGN:
Intervention Model Description: prospective, single arm, un-blinded, multi-center early feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Device Implantation (Experimental): To epicardially reshape the mitral valve annulus and left ventricle without the need for cardiopulmonary bypass (CPB) and open-heart access (atriotomy) using an epicardial implant.
  Interventions: Device: Implant an epicardial device to reshape the mitral valve annulus

INTERVENTIONS:
Device: Implant an epicardial device to reshape the mitral valve annulus — The implant is intended to epicardially reshape the mitral valve annulus and left ventricle without the need for cardiopulmonary bypass (CPB) and open-heart access (atriotomy), in patients with left ventricular dilation and mitral valve insufficiency in patients with ischemic or functional MR.

SUMMARY:
To evaluate the safety and performance of the Mitral Touch System to treat mitral insufficiency in patients who are to undergo cardiac surgery with either a sternotomy or thoracotomy who present with moderate to severe ischemic or functional mitral regurgitation.

DETAILED DESCRIPTION:
The Mitral Touch Systems is intended to epicardially reshape the mitral valve annulus and left ventricle without the need for cardiopulmonary bypass (CPB) and open-heart access (atriotomy), in patients with left ventricular dilation and mitral valve insufficiency in patients with ischemic or functional MR.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or greater (2+) ischemic
* Functional Mitral regurgitation by 2D echocardiography using an integrative method
* Patient is scheduled for cardiac surgery (e.g. CABG including patients on the waiting list for Heart Transplantation)
* Patient is 22 years of age or older
* Patient is willing and able to sign Informed Consent Form
* Within 90 days patients should be on stable optimally uptitrated medical therapy recommended according to current guidelines23 as standard of care for heart failure therapy in the United States

Exclusion Criteria:

* Any evidence of structural (chordal or leaflet) mitral valve disease
* Inability to derive ERO, LVESVI or LVEDVI by TTE
* Prior surgical or percutaneous mitral valve intervention
* Contraindication to cardiopulmonary bypass (CPB)
* Clinical signs of cardiogenic shock
* Treatment with chronic intravenous inotropic therapy
* Severe, irreversible pulmonary hypertension in the judgement of the investigator
* ST segment elevation requiring intervention within 7 days prior to randomization
* Congenital heart disease (except PFO or ASD)
* Evidence of cirrhosis or hepatic synthetic failure
* Renal insufficiency (eGFR < 30 ml/min)
* History of endocarditis or current endocarditis
* Ejection fraction <25%
* NY heart class IV
* MV diameters > 7cm
* Any coronary artery calcification at site of placement as determined by angiogram
* Myxomatous mitral regurgitation
* Women who are pregnant (by history of menstrual period or pregnancy test if history is considered unreliable)
* Abnormal cardiac anatomy discovered prior to surgery or during procedure
* Pericardial adhesions
* Insufficient clinical signature reduction of mitral regurgitation during device sizing and placement. (No device remains, patient moved to only 30-Day follow-up.)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-10 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Freedom from Major Adverse Events | Procedure through 30 days
  Freedom from Major Adverse Events such as death, stroke, Increase of NYHA >1, Re-Hospitalization or reoperation of the Mitral Valve

SECONDARY OUTCOMES:
Rate of Technical Feasibility to implant the Mitral Touch Device | Procedure
  Septal lateral diameter reduction of the mitral valve at implantation, Reduction in MR Grade by at least 1 grade from baseline
Rate of Freedom from Serious Adverse Events from Implantation of the Mitral Touch Device | procedure
  Implantation of the Mitral Touch Device without Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Smith II, MD, Principal Investigator — Baylor Scott and White Medical Center
Locations (1):
- Baylor Scott and White, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No